CLINICAL TRIAL: NCT05377866
Title: Holo CTO Proctoring Study
Status: Completed | Type: Observational
Sponsor: Sorlandet Hospital HF (Other Government)
Collaborators: Oslo University Hospital (Other); HoloCare AS (Industry)
Responsible Party: Sponsor
Other Study IDs: HoloCTO
Record Dates: First submitted 2021-09-27; First posted 2022-05-17 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2021-09

CONDITIONS: Percutaneous Coronary Intervention; Chronic Total Occlusion of Coronary Artery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study population: Patients undergoing percutaneus coronary intervention for chronic total occlusion. The procedures will all be done using mixed reality to enable remote proctoring. The study is a feasibility trial.
  Interventions: Other: Remote proctoring using HoloLens

INTERVENTIONS:
Other: Remote proctoring using HoloLens — Assess Microsoft HoloLens as an interactive communication device in remote proctoring, and enhancement of teamwork in complex CTO procedures.
  Other Names: Chronic total occlusion percutaneus coronary intervention

SUMMARY:
Assess Microsoft HoloLens as an interactive communication device in remote proctoring, and enhancement of teamwork in complex CTO procedures

DETAILED DESCRIPTION:
Proctoring in medicine is related to better outcomes. Specifically, in CTO PCI systematic proctoring has demonstrated improved success rates, and an increased ability to treat lesions that are more complex. Most likely, proctoring together with operator volume is one of the foundations to the introduction and execution of CTO procedures. Proctoring traditionally involves an expert operator (proctor), visiting the institution, performing the procedure together with the local operator. This involves increased cost, and current travel restrictions makes traditional one-on-one proctoring challenging.

This study aims to evaluate the Microsoft HoloLens as a potential platform in proctoring and effective real time communication between PCI operators located at different geographical locations. The proctor and the local operator interact using a head mounted mixed reality (MR) display, enabling the proctor to see the same image as the operator, from any distanced location.

ELIGIBILITY:
Inclusion Criteria:

Clinical inclusion criteria:

* Stable angina pectoris, or dyspnoea as an angina equivalent
* Age ≥18 yrs.
* Able to provide written informed consent

Angiographic inclusion criteria:

* One or more completely occluded coronary arteries with Thrombolysis In Myocardial Infarction (TIMI) flow 0. An estimated occlusion duration of at least 3 months
* Absence of Q-wave in ECG leads corresponding to the occluded vessel, or documented viability of the main territory by MRI or echocardiography

Procedural inclusion criteria:

* Clinical indication for CTO PCI regardless of operative technique

Exclusion Criteria:

* STEMI within 72 hours
* Cardiogenic shock
* Active bleeding or coagulopathy
* Life expectancy < 2 years
* Relevant allergies (aspirin, clopidrogrel, ticagrelol, contrast compounds)
* Severe peripheral artery disease
* Clinical unstable angina

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary artery disease and total chronic occlusion of one or more coronary arteries.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2021-11-04 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Standard Usability Score on a Likert Scale | Procedure duration( aprox 120 min)
  The operators completing the intervention will rate the usability of the system on a Likert scale:
  1. The HoloLens was useful in this procedure
  2. The HoloLens was not distracting
  3. The HoloLens was comfortable to wear
  4. The HoloLens camera image has sufficient quality for clinical use (not considering the fluoroscopy screen)
  5. Compared to an alternative system with fluoroscopy image plus handsfree voice (telephone), the HoloLens gives additional value during the procedure
  6. The current solution with Remote Assist plus parallel fluoroscopy streaming is mature enough for routine use
  7. The current solution is stable
  8. The current solution is easy to set up prior to the procedure
  9. I would like to continue to use the HoloLens in CTO procedures routinely when remote proctoring is needed
  Agree to Disagree Likert Scale
  * Strongly Disagree
  * Disagree
  * Neither agree nor disagree
  * Agree
  * Strongly Agree

CONTACTS AND LOCATIONS:
Overall Officials: Slobodan Calic, MD, Principal Investigator — Sorlandet Hospital
Locations (1):
- Sorlandet Hospital, Arendal, Agder, Norway

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2021-10-17): https://cdn.clinicaltrials.gov/large-docs/66/NCT05377866/Prot_000.pdf